CLINICAL TRIAL: NCT04567524
Title: A Multiple Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of Risperidone Extended Release Capsules in Subjects With Schizophrenia, Schizoaffective Disorder
Brief Title: A Multiple Dose Study to Assess the Safety, Tolerability and PK of Risperidone Extended Release Capsules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lyndra Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYN-005-C-004
Record Dates: First submitted 2020-09-16; First posted 2020-09-28 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia Schizoaffective
MeSH Terms: conditions — Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Intervention Model Description: LYN-005-C-004 was a blinded, multiple-dose, randomized, parallel group, safety, tolerability and PK study of LYN-005 in subjects with a primary diagnosis of schizophrenia or schizoaffective disorder in general good health. Eligible subjects were clinically stable and receiving a therapeutic dose of an approved oral antipsychotic drug for a minimum of 6 weeks at the time of Screening. Enrolled subjects were evaluated under steady-state conditions on commercially-available IR risperidone tablets and then assigned in blinded fashion either to LYN-005 weekly or continued encapsulated IR risperidone daily for 3 weeks to attain (or continue) steady-state exposure.
Who Masked: Participant, Care Provider
Masking Description: Although treatment assignment was blinded; the dose level was not blinded. The dose of LYN-005 (14 or 28 mg)/IR risperidone (2 or 4 mg/day) administered was based on the subject's current antipsychotic medication dose. Randomization was stratified by risperidone dose (LYN-005 14 mg/IR risperidone 2 mg/day [low dose] and LYN-005 28 mg/IR risperidone 4 mg/day [high dose], with a maximum of 16 subjects enrolled in each stratum. Within each stratum, subjects were randomized on a 3:1 basis to either LYN-005 or risperidone, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): LYN-005: capsules containing LYN-005 stellate; the 14mg dose of LYN-005 contains 3 active arms containing risperidone, and 3 inactive arms and the 28 mg dose of LYN-005 contains 6 active arms containing risperidone.
  AND
  IR Risperidone Matched Placebo: Orange capsule-shaped tablets containing inactive ingredient.
  Interventions: Drug: LYN-005
- Arm 2 (Placebo Comparator): LYN-005 Matched Placebo: Size 00EL capsules containing inactive ingredient with no stellate.
  AND
  IR Risperidone: Risperidone 2 mg (orange) capsule-shaped tablets.
  Interventions: Drug: LYN-005

INTERVENTIONS:
Drug: LYN-005 — LYN-005 (14 or 28 mg weekly) plus IR risperidone matched placebo.
  Other Names: Risperidone

SUMMARY:
Lyndra is developing an oral, extended release (ER) formulation of risperidone (LYN-005) presented in a capsule dosage form with the intent of reducing the frequency of dosing orally-administered medications to once weekly or less and thereby improving the management of schizophrenia.

Study LYN-005-C-004 will evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple dose administration of the ER formulation at two dose levels of LYN-005 relative to IR risperidone.

DETAILED DESCRIPTION:
LYN-005-C-004 is a blinded, multiple-dose, randomized, parallel group, safety, tolerability and PK study of LYN-005 in subjects with a primary diagnosis of schizophrenia or schizoaffective disorder in general good health. Eligible subjects must be clinically stable and receiving a therapeutic dose of an approved oral antipsychotic drug for a minimum of 6 weeks at the time of Screening. Enrolled subjects will be evaluated under steady-state conditions on commercially-available IR risperidone tablets and then assigned in blinded fashion either to LYN-005 weekly or continued encapsulated IR risperidone daily for 3 weeks to attain (or continue) steady-state exposure.

ELIGIBILITY:
Inclusion Criteria: Eligibility for this study was met if each one of the following inclusion criteria was satisfied at Screening (or at baseline when specified):

1. Male or female aged ≥18 and ≤50 years.
2. Current diagnosis of schizophrenia or schizoaffective disorder according to DSM-5 criteria as confirmed by the MINI 7.0.2.
3. The following psychiatric criteria were used to determine subject eligibility:

   1. Duration of diagnosis of schizophrenia or schizoaffective disorder of ≥2 years.
   2. Outpatient; not hospitalized for worsening of schizophrenia within the last 6 months (partial hospitalization for social management within this time period is acceptable).
   3. Medically stable over the last month and psychiatrically stable without significant symptom exacerbation over the last 3 months.
4. Stabilized on an oral antipsychotic medication (single agent) for a minimum of 6 weeks at the time of Screening.
5. On a stable dosage of all permitted non-antipsychotic medications (except for medication to be used on an as-needed basis) for at least 1 month prior to the Screening visit and for the duration of the study.
6. CGI-S score of ≤4 (moderately ill).
7. PANSS score of ≤80 points.
8. Body mass index (BMI) of ≥18 kg/m2 and ≤35 kg/m2.
9. Able to read and understand study procedures and provide written informed consent before the initiation of any protocol-specific procedures.
10. Willing to comply with all protocol-specified procedures and availability for the duration of the study.
11. Subject has identified a caregiver or personal contact with whom the subject communicates with at least once a week.

Exclusion Criteria: Subject will not be considered eligible to participate in this study if any one of the following exclusion criteria is satisfied at Screening (or at baseline when specified):

1. Subjects with known clinically significant esophageal or GI disease, including but not limited to:

   1. Known strictures such as esophageal web, pyloric stenosis, or small intestinal stricture, or subjects with high risk of stricture, e.g., Crohn's disease.
   2. Diagnosis of a condition known to elevate or lower gastric pH, e.g., achlorhydria or hypochlorhydria.
   3. Prior varices or small or large bowel obstructions.
   4. Prior abdominal or upper gastrointestinal surgery (prior uncomplicated laparoscopic procedures including appendectomy or colectomy).
   5. History of dysphagia or aspiration in the last 5 years.
   6. History of an esophageal motility disorder or undergoing treatment for a gastric motility disorder.
   7. Significant history of diarrhea or constipation within 3 months of Screening
   8. Multiple episodes of abdominal pain within 3 months of Screening.
   9. Subjects who experience moderate or severe dysmenorrhea or menorrhagia (with use of pain medication) within 3 months of Screening.
   10. History of moderate to severe Acid Reflux Disease or a score of ≥2 on the Acid Reflux Severity Scale (ARSS) [2], indicating moderate to severe symptoms. The ARSS scale is as follows:

   None = 0 no symptoms Mild = 1 awareness of symptom, but easily tolerated Moderate = 2 discomfort sufficient to cause interference with normal activities Severe = 3 incapacitating, with inability to perform normal activities.
2. Subjects with PILL-5 questionnaire score of 5 or greater.
3. Medical history or current diagnoses indicating the presence of any of the below conditions:

   1. Presence of an uncontrolled, unstable, clinically significant medical condition could that could put the subject at risk because of participation in the study, interfere with the subject's ability to participate in the study or influence the interpretation of safety or PK evaluations.
   2. History of a major cardiovascular event (myocardial infarction, cardiac surgery or revascularization, unstable angina, stroke, or transient ischemic attack) or a hospitalization for heart failure with 6 months of Screening.
   3. Any clinically significant illness, medical or surgical procedure or trauma within 4 weeks of Screening.
   4. Known immunocompromised status, including individuals who have undergone organ transplantation, on immunosuppression for an immunemediated disease, or are positive for human immunodeficiency virus (HIV).
   5. Subjects with a positive test for active hepatitis B or C at Screening. Subjects with successfully treated hepatitis B infection which has been resolved for greater than 1 year or successfully treated hepatitis C infection will not be excluded.
   6. Subjects who have donated more than 250 mL of blood within 30 days of Screening.
   7. Subjects who have difficulties with venipuncture/cannulation, including difficulty accessing veins for blood sampling and/or history of coagulopathy or endocarditis.
   8. Subjects with a current DSM-5 diagnosis of major depressive episode, panic disorder, agoraphobia, social anxiety disorder, obsessive- compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder on the MINI 7.0.2 or in the judgment of the Investigator. (Note that individuals with depression secondary to schizoaffective disorder are eligible).
   9. Suicidal ideation associated with actual intent and a method or plan in the past 6 months, as measured by the C-SSRS (i.e., "Yes" answers on items 4 or 5) at Screening or having made a suicide attempt within the last 2 years.
   10. Known or suspected (non-febrile) seizure disorder.
   11. History of neuroleptic malignant syndrome.
   12. Current or history of clinically significant tardive dyskinesia.
   13. Known or suspected diagnosis of intellectual disability or organic brain disorder or other diagnosis that is primarily responsible for current symptoms and functional impairment.
   14. Medically non-adherent in the management of their schizophrenia/schizoaffective disorder.
4. Use of the below medications/treatments in the 2 weeks before enrollment, including:

   1. Proton pump inhibitors or H2 blockers.
   2. Prokinetic agents.
   3. Medications that may interfere with the absorption, metabolism, or excretion of risperidone, e.g.:

      Drugs metabolized via CYP3A4 pathway, such as macrolide antibiotics and azole antifungals). Moderate or strong CYP3A4 p-glycoprotein (P-gp) enzyme inducers and inhibitors (carbamazepine, phenytoin, rifampicin, phenobarbital, itraconazole, verapamil). Moderate or strong CYP2D6 inhibitors (e.g., fluoxetine, fluoxetine combinations, paroxetine), or quinidine.
   4. Concomitant medications, natural remedies, supplements or vitamins which are associated with changes to gastric motility or pH. Use of antacids is permissible, except within 2 hours of dosing with LYN-005.
   5. Benzodiazepines; except lorazepam, diazepam and oxazepam, which are acceptable if for the treatment of depression, anxiety or insomnia.
   6. Use of more than one antidepressant; or if on just one, a change in dose within 6 weeks of Screening.
   7. Depot antipsychotic use within 9 months of Screening.
   8. Electroconvulsive therapy within 3 months of Screening.
5. Subjects with clinically significant abnormal safety (e.g. physical examination, vital sign) or safety laboratory assessments, specifically:

   1. Presence of a clinically significant abnormal laboratory result on blood or urine safety tests at Screening.
   2. Anemia (hemoglobin below lower limit of normal reference range) at Screening.
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≥3.0 × upper limit of normal (ULN), or total bilirubin ≥1.5 × ULN.
   4. Moderate or severe renal insufficiency at Screening (glomerular filtration rate <60 mL/min, as determined using the Cockcroft-Gault formula).
   5. Heart rate of <50 beats per minute (bpm) at Screening.
   6. Systolic blood pressure ≤100 or ≥150 and/or diastolic blood pressure ≤60 mmgHg or ≥100 mmHg at Screening.
   7. HbA1c ≥6.5% at Screening.
   8. Positive fecal occult blood test at Screening
   9. Clinically significant prolactin elevation (≥200 ng/mL for females; ≥100 ng/mL for males).
6. Subjects with the below specified patterns of substance use at Screening:

   1. Fulfillment of the DSM-5 criteria for moderate or severe substance use disorder (excluding nicotine and caffeine) within 6 months of Screening.
   2. History of alcohol consumption exceeding moderate use; in males exceeding 21 units per week and in females exceeding 14 units per week (1 unit = 360 ml beer, 25 mL of 40% spirit or a 125 mL glass of wine) over the past month. Subjects are not permitted to consume alcohol during the inpatient stay nor 12 hours before any clinic visit while outpatient.
   3. Positive ethanol breathalyzer.
   4. Positive urine drug screen for substances of abuse other than cannabis.
   5. Heavy nicotine use (consumption of >40 cigarettes or >36 mg of nicotine from other sources [e.g., vaping products] daily) or daily use of smokeless tobacco.
7. Subjects of reproductive potential who are (hetero) sexually active but unwilling to use acceptable means of contraception through the EOS. For clarity, subjects who are at least 1 year post-menopausal are not of reproductive potential. Acceptable means of contraception include:

   1. Subjects who have been surgically sterilized.
   2. Females of reproductive potential: diaphragm, injectable, oral/patch contraceptives for a minimum of 6 weeks, contraceptive sponge, implant, or intrauterine device in use prior to enrollment.
   3. Males: condom in combination with any of the above means of contraception.
   4. All subjects: abstinence may be an acceptable means of contraception as long as the individual consents to initiate immediate use of double barrier protection for the duration of the study should (hetero) sexual intercourse occur.
8. Subjects who are nursing or who have positive or indeterminate pregnancy tests at either Screening (serum test) or enrollment (urine test).
9. Use of any experimental agent within 1 month or 5 half-lives of Screening, whichever is longer.
10. Subjects who are employees or immediate family members of employees of the site, Sponsor or study-related vendors.
11. History of a serious allergic or hypersensitivity reaction to risperidone or LYN-005 excipients (refer to Investigator's Brochure).
12. Subjects with history of X-ray, computed tomography (CT) scan or angiogram of the abdomen within one year of Screening.
13. Subjects with CYP2D6 poor or underdetermined metabolizer status based on genetic testing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Scranton, MD, MPH, Principal Investigator — Chief Medical Officer
Locations (5):
- United States (5):
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Hassman Research Institute, Marlton, New Jersey
  - Community Clinical Research, Inc, Austin, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites that randomized participants in the US. The study period was 13 August 2020 (first signed informed consent) to 22 December 2020 (last participant visit/observation)
Pre-assignment Details: A total of 34 participants were enrolled. Thirty-two participants completed the Run-in Period and were randomized, comprising the Safety Population; of these, 24 participants received LYN-005 (12 low dose; 12 high dose) and 8 participants received IR risperidone (4 low dose; 4 high dose).
Groups:
- LYN-005 14mg: LYN-005: Size 00EL capsules containing LYN-005 stellate (14mg)
  AND
  IR risperidone matched placebo
- LYN-005 28mg: LYN-005: Size 00EL capsules containing LYN-005 stellate (28 mg)
  AND
  IR risperidone matched placebo
- Risperidone 2 mg: Risperidone (2 mg)
  AND
  LYN-005-matched placebo
- Risperidone 4 mg: Risperidone (4 mg)
  AND
  LYN-005-matched placebo.
Period: Overall Study
Arm/Group | LYN-005 14mg | LYN-005 28mg | Risperidone 2 mg | Risperidone 4 mg
Started | 12 | 12 | 4 | 4
Completed | 9 | 11 | 4 | 3
Not Completed | 3 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- LYN-005 14 mg: LYN-005: Size 00EL capsules containing LYN-005 stellate (14mg)
  AND
  IR risperidone matched placebo
- LYN-005 28 mg: LYN-005: Size 00EL capsules containing LYN-005 stellate (28 mg)
  AND
  IR risperidone matched placebo
- Total: Total of all reporting groups
Arm/Group | LYN-005 14 mg | LYN-005 28 mg | Risperidone 2 mg | Risperidone 4 mg | Total
Number analyzed (Participants) | 12 | 12 | 4 | 4 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (6.24) | 34.3 (7.46) | 35.0 (7.12) | 43.5 (7.85) | 36.2 (7.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 0 | 6
  Male | 10 | 9 | 3 | 4 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 11 | 11 | 4 | 4 | 30
  Race: White | 1 | 1 | 0 | 0 | 2
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.57 (4.695) | 24.98 (4.476) | 26.48 (2.680) | 26.78 (6.086) | 27.11 (4.835)
ESRS Total Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — ESRS = Extrapyramidal Symptom Rating Scale Extrapyramidal Symptom Rating Scale (ESRS) was developed to assess four types of drug-induced movement disorders (DIMD): Parkinsonism, akathisia, dystonia, and tardive dyskinesia (TD). The range of this scale is 0 to 25.
  An increase in ESRS score indicates a worse outcome.
  units on a scale | 0.2 (0.58) | 0.6 (2.02) | 0 (0) | 0.8 (1.5) | 0.4 (1.36)
CGI-S Total Score at Baseline [Mean (Standard Deviation); unit: units on a scale] — CGI-S = Clinical Global Impression - Severity The CGI rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with psychiatric disorders. CGI-S is a scale (1 to 7).
  An increase in CGI-S score indicates a worse outcome
  units on a scale | 2.9 (0.51) | 3.0 (0.85) | 2.8 (0.50) | 3.3 (0.50) | 3.0 (0.65)

OUTCOME MEASURES:

1. Primary Outcome: Participants With at Least One Treatment Emergent Adverse Event (TEAE).
Description: Incidence of treatment emergent adverse events (TEAEs) reported as participants with at least one treatment emergent adverse event (TEAE).
Time Frame: 35 days
Population: Safety Population: All enrolled participants who were randomized to study drug (LYN-005 14 mg/28 mg or IR risperidone 2 mg/4 mg) and received at least 1 dose of randomized study drug. Participants were reported according to the treatment received. The Safety Population was the primary safety analysis population.
Measure: Number; unit: Number of Participants with TEAEs
Groups:
- Overall LYN-005: LYN-005 (14 mg) + LYN-005 (28 mg)
- Overall Risperidone: Risperidone (2 mg) + Risperidone (4 mg)
Arm/Group | LYN-005 14mg | LYN-005 28mg | Overall LYN-005 | Risperidone 2 mg | Risperidone 4 mg | Overall Risperidone
Number analyzed (Participants) | 12 | 12 | 24 | 4 | 4 | 8
Number of Participants with TEAEs | 10 | 8 | 18 | 1 | 1 | 2

2. Primary Outcome: Total Number of Treatment Emergent Adverse Events (TEAEs).
Description: Incidence of treatment emergent adverse events (TEAEs) reported as total number of TEAEs.
Time Frame: 35 days
Population: as for outcome 1
Measure: Number; unit: Number of Experienced TEAEs
Arm/Group | LYN-005 14mg | LYN-005 28mg | Overall LYN-005 | Risperidone 2 mg | Risperidone 4 mg | Overall Risperidone
Number analyzed (Participants) | 12 | 12 | 24 | 4 | 4 | 8
Number of Experienced TEAEs | 15 | 21 | 36 | 2 | 2 | 4

3. Primary Outcome: Active Moiety PK (Cmax)
Description: Active moiety Cmax (risperidone and 9-hydroxyrisperidone combined) after repeat weekly doses of LYN-005 Extended Release (ER) capsules relative to Immediate Release (IR) risperidone tablets at 2 dose levels.
Time Frame: Reported data was obtained following multiple dose administration of 3 weekly doses [(IR, Day-1), (ER, Week 1), ER Week 3)] of 14 or 28 mg risperidone LYN-005 capsules to assess extended release PK.
Population: All enrolled participants who received at least 1 dose of randomized study drug and had at least 1 post-dose quantifiable (or evaluable) PK concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- LYN-005 14 mg (A): 2 mg Risperidone to 14 mg LYN-005 (IR, Day -1)
- LYN-005 14 mg (B): 2 mg Risperidone to 14 mg LYN-005 (ER, Week 1)
- LYN-005 14 mg (C): 2 mg Risperidone to 14 mg LYN-005 (ER, Week 3)
- Risperidone 2 mg (A): 2 mg Risperidone to 2 mg Risperidone (IR, Day -1)
- Risperidone 2 mg (B): 2 mg Risperidone to 2 mg Risperidone (IR, Day 1)
- Risperidone 2 mg (C): 2 mg Risperidone to 2 mg Risperidone (IR, Day 15)
- LYN-005 28 mg (A): 4 mg Risperidone to 28 mg LYN-005 (IR, Day -1)
- LYN-005 28 mg (B): 4 mg Risperidone to 28 mg LYN-005 (ER, Week 1)
- LYN-005 28 mg (C): 4 mg Risperidone to 28 mg LYN-005 (ER, Week 3)
- Risperidone 4 mg (A): 4 mg Risperidone to 4 mg Risperidone (IR, Day -1)
- Risperidone 4 mg (B): 4 mg Risperidone to 4 mg Risperidone (IR, Day 1)
- Risperidone 4 mg (C): 4 mg Risperidone to 4 mg Risperidone (IR, Day 15)
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 12 | 12 | 11 | 4 | 4 | 3
ng/mL | 31.0 (37.5) | 20.0 (56.7) | 18.6 (42.9) | 24.8 (38.3) | 30.3 (17.5) | 31.2 (68.7) | 24.6 (405.7) | 31.2 (32.1) | 30.4 (102.7) | 54.1 (19.3) | 46.3 (23.8) | 48.8 (40.9)

4. Primary Outcome: Active Moiety PK (AUC0-24, AUC0-168)
Description: Active moiety AUC (risperidone and 9-hydroxyrisperidone combined) after repeat weekly doses of LYN-005 ER capsules relative to IR risperidone tablets at 2 dose levels.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- LYN-005 14 mg (C): 2 mg Risperidone to 14 mg LYN-005 (ER Week 3)
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 12 | 12 | 11 | 4 | 4 | 3
h*ng/mL
  AUC0-24 | 377 (44.0) | 361 (49.0) | 371 (47.4) | 301 (23.1) | 326 (19.1) | 359 (32.6) | 472 (137.7) | 575 (39.3) | 568 (104.3) | 732 (46.3) | 753 (44.9) | 687 (36.9)
  AUC0-168: number analyzed (Participants) | 0 | 12 | 11 | 0 | 0 | 0 | 0 | 12 | 11 | 0 | 0 | 0
  AUC0-168 |  | 1820 (52.1) | 2120 (53.2) |  |  |  |  | 3350 (42.3) | 2950 (121.1) |  |  |

5. Primary Outcome: Active Moiety Tmax
Description: Active Moiety Tmax (h) (risperidone and 9-hydroxyrisperidone combined) after repeat weekly doses of LYN-005 ER capsules relative to IR risperidone tablets at 2 dose levels.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 12 | 12 | 11 | 4 | 4 | 3
hours | 1.9 [0.0 to 4.0] | 23.7 [4.0 to 120.0] | 23.8 [0.0 to 72.0] | 3.0 [1.0 to 4.0] | 1.5 [1.0 to 2.0] | 3.0 [2.0 to 4.0] | 1.0 [0.6 to 7.9] | 24.1 [6.1 to 72.5] | 23.8 [0.0 to 169.0] | 2.1 [0.8 to 6.0] | 4.0 [1.1 to 6.1] | 2.0 [2.0 to 2.1]

6. Secondary Outcome: PK of Risperidone (Cmax).
Description: To characterize exposure (Cmax) of risperidone during the switch to LYN-005.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 12 | 12 | 11 | 4 | 4 | 3
ng/mL | 11.7 (58.2) | 4.44 (95.3) | 4.07 (59.1) | 9.97 (111.0) | 12.3 (40.5) | 15.6 (84.2) | 21.2 (55.6) | 6.87 (72.7) | 7.39 (230.9) | 17.0 (21.2) | 13.5 (32.6) | 14.0 (33.0)

7. Secondary Outcome: PK of Risperidone (AUC0-24h, AUC0-168).
Description: To characterize exposure (AUC0-24h, AUC0-168) of risperidone during the switch to LYN-005.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 12 | 12 | 11 | 4 | 4 | 3
h*ng/mL
  AUC0-24h | 54.9 (81.5) | 65.8 (93.3) | 65.2 (66.6) | 43.4 (131.2) | 47.7 (103.5) | 86.2 (58.1) | 113 (109.9) | 111 (88.1) | 119 (257.4) | 87.1 (67.2) | 82.4 (67.0) | 84.4 (80.5)
  AUC0-168: number analyzed (Participants) | 0 | 12 | 11 | 0 | 0 | 0 | 0 | 12 | 11 | 0 | 0 | 0
  AUC0-168 |  | 227 (87.3) | 306 (67.1) |  |  |  |  | 806 (91.2) | 453 (276.8) |  |  |

8. Secondary Outcome: PK of 9-Hydroxyrisperidone (Cmax).
Description: To characterize exposure (Cmax) of 9-Hydroxyrisperidone during the switch to LYN-005.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 11 | 12 | 11 | 4 | 4 | 3
ng/mL | 20.8 (31.0) | 16.1 (49.6) | 15.6 (41.9) | 15.5 (12.1) | 17.5 (37.8) | 16.9 (53.3) | 16.0 (282.3) | 24.7 (26.0) | 22.5 (91.1) | 39.6 (22.9) | 35.7 (24.5) | 36.2 (38.4)

9. Secondary Outcome: PK of 9-Hydroxyrisperidone (AUC0-24h, AUC0-168h).
Description: To characterize exposure (AUC0-24h, AUC0-168h) of 9-Hydroxyrisperidone during the switch to LYN-005.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | LYN-005 14 mg (A) | LYN-005 14 mg (B) | LYN-005 14 mg (C) | Risperidone 2 mg (A) | Risperidone 2 mg (B) | Risperidone 2 mg (C) | LYN-005 28 mg (A) | LYN-005 28 mg (B) | LYN-005 28 mg (C) | Risperidone 4 mg (A) | Risperidone 4 mg (B) | Risperidone 4 mg (C)
Number analyzed (Participants) | 12 | 12 | 11 | 4 | 4 | 4 | 11 | 12 | 11 | 4 | 4 | 3
h*ng/mL
  AUC0-24h | 315 (39.7) | 268 (38.2) | 302 (47.0) | 243 (11.2) | 262 (20.8) | 265 (26.6) | 268 (272.6) | 441 (33.6) | 523 (177.9) | 641 (43.5) | 665 (42.9) | 645 (45.5)
  AUC0-168h: number analyzed (Participants) | 0 | 12 | 11 | 0 | 0 | 0 | 0 | 12 | 11 | 0 | 0 | 0
  AUC0-168h |  | 1530 (51.7) | 1770 (54.4) |  |  |  |  | 2720 (35.9) | 2090 (100.5) |  |  |

ADVERSE EVENTS:
Time Frame: 35 days Double-blind Period consisted of the period between Day 1 to Day 35.
Description: Safety Population consisted of all enrolled participants who were randomized to study drug (LYN-005 Low/High: 14 mg/28 mg or IR Risperidone Low/High: 2 mg/4 mg) and received at least 1 dose of randomized study drug. Double-blind Period consisted of the period between Day 1 to Day 35. If a participant had multiple AEs meeting a definition, the participant was presented only once in the respective participant count [n (%)].
Groups:
- IR Risperidone 2 mg: Risperidone (2 mg)
  AND
  LYN-005-matched placebo
- IR Risperidone 4 mg: Risperidone (4 mg)
  AND
  LYN-005-matched placebo.
Arm/Group | LYN-005 14 mg | LYN-005 28 mg | IR Risperidone 2 mg | IR Risperidone 4 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 10/12 | 8/12 | 1/4 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYN-005 14 mg (N=12) | LYN-005 28 mg (N=12) | IR Risperidone 2 mg (N=4) | IR Risperidone 4 mg (N=4)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occult Blood Positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Akathisia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperprolactinaemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT04567524/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04567524/SAP_003.pdf